CLINICAL TRIAL: NCT00160901
Title: Prospective Randomized Trial With Complementary Therapies During Chemotherapy at the Women's Hospital of the University of Heidelberg
Brief Title: Complementary Therapies for the Reduction of Side Effects During Chemotherapy for Breast Cancer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Heidelberg University (Other)
Collaborators: Hector-Stiftung (Other); Cefak KG, Kempten (Unknown); Ursapharm, Saarbrücken (Unknown); Schwabe-Wenex International Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M16
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2007-04-19 (Estimated); Status verified 2007-03

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Chemotherapy; Phytotherapy; Nutritional counseling
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: two complex naturopathic add-on therapies, leaflet 5-a-day

SUMMARY:
The purpose of this study is to determine wether a complementary therapy consisting of a combined medication of selenium, milk thistle, goldenrod and bromelain and a consultation concerning nutrition and physical activity can reduce side effects of a chemotherapy in breast cancer patients.

DETAILED DESCRIPTION:
patients were randomized to receive: (a) individual nutrition consultation with recommendations for physical activity before or on the first day of chemotherapy together with daily oral medication consisting of selenium (sodium-selenit 100 microg/d), milk thistle (silibin 280 mg/d), goldenrod (solidago 1,680g/d) and pineapple enzyme (bromelaine 3.000 F.I.P. units/d) during the first three cycles till 3-5 weeks later, (b) individual nutrition consultation with recommendations for physical activity only and (c) a leaflet "5-a-day" for the control group.

Primary endpoint was the difference of the global health status from the EORTC QLQ-C30 before and 3-5 weeks after the third cycle of chemotherapy. Secondary endpoints were the other subscales of the EORTC QLQ C3o and BR 23 and anxiety and depression from the HADS-D.

ELIGIBILITY:
Inclusion Criteria:

* Indication for chemotherapy for breast cancer for at least 3 cycles

Exclusion Criteria:

* Prior chemotherapy within 12 months
* use of herbal or nutritional supplements or other complementary or alternative medications ≥ 7 days prior to start of chemotherapy and during the trial
* allergy to study medication
* Selenium intoxication
* Current use of cumarins or other medication influencing the coagulation system
* Edema in case of impaired cardial or renal function
* Other severe medical condition
* Psychiatric or central neurological disorders
* Regular fluid intake < 2000 ml per day

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2003-08; Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Difference in the sum score of the most common side effects of a chemotherapy (fatigue, nausea, loss of appetite, constipation, diarrhea) measured by the EORTC QLQ C30 3-5 weeks after and before 3 cycles of chemotherapy

SECONDARY OUTCOMES:
Difference in general QOL 3-5 weeks after and before three cycles of chemotherapy
Difference in anxiety and depression measured by HADS-D 3-5 weeks after and before three cycles of chemotherapy
Sensitivities measured by the perimed sensitivity questionnaire
Creatinin
ALAT
Coagulation time
Selenium

CONTACTS AND LOCATIONS:
Overall Officials: Cornelia U. von Hagens, MD, Principal Investigator — Department of Complementary and Integrative Medicine Women's Hospital, University of Heidelberg
Locations (1):
- Department of Complementary and Integrative Medicine, Heidelberg, Baden-Wurttemberg, Germany